CLINICAL TRIAL: NCT03628729
Title: Investigation of the Incidence of Caries in Pits and Fissures Sealed With Bioactive Sealant
Brief Title: Investigation of the Incidence of Caries in Pits and Fissures Sealed With Bioactive Sealant Compared to Fluoride Releasing Resin Based Pit and Fissure Sealant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed tarek heiba, Master student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CEBD-CU-2018-07-17
Record Dates: First submitted 2018-07-25; First posted 2018-08-14 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Pit and Fissure Caries
MeSH Terms: conditions — Van der Woude syndrome | interventions — Pit and Fissure Sealants

STUDY DESIGN:
Intervention Model Description: A total of 40 volunteer patients with at least 2 non-cavitated molar teeth will be assigned in this study. Patients will be randomly divided into two groups according to type of sealant (S) where in group S1, pits and fissures will be sealed with bioactive pits-and-fissure sealant; while group S2, pits and fissures will be sealed with fluoride releasing resin based pits and fissures sealant. Each restoration will be assessed after three, six months.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embrace™ WetBond™ Pit & Fissure Sealant. (Experimental): pits and fissures will be sealed with bioactive pits-and-fissure sealant
  Interventions: Other: Embrace™ WetBond™ Pit & Fissure Sealant
- Seal-Rite™ Pit & Fissure Sealant, Pulpdent Corportation, USA (Active Comparator): Pits and fissures will be sealed by fluoride releasing resin based pits and fissures sealant
  Interventions: Other: Seal-Rite™ Pit & Fissure Sealant, Pulpdent Corportation, USA

INTERVENTIONS:
Other: Embrace™ WetBond™ Pit & Fissure Sealant — pit and fissure sealant that contain the precursor in the formation of hydroxyapatite which is Amorphous Calcium Phosphate (ACP) ,which has anti-cariogenic effect as well as remineralization potential as it contain bioactive material which stimulate crystal growth within the lesion by increasing the concentration of calcium and phosphate ions
  Arms: Embrace™ WetBond™ Pit & Fissure Sealant.
Other: Seal-Rite™ Pit & Fissure Sealant, Pulpdent Corportation, USA — Fluoride releasing resin based pits and fissures sealant
  Arms: Seal-Rite™ Pit & Fissure Sealant, Pulpdent Corportation, USA

SUMMARY:
This study will be conducted to investigate the incidence of caries in pits and fissures sealed with a bioactive sealant compared to a fluoride releasing resin based pits and fissures sealant in preventive treatment procedures in adult population over a six months period.

DETAILED DESCRIPTION:
The study will be conducted in Conservative Dentistry Department, Faculty of Dentistry, Cairo University, The operator in charge will be: Mohamed Tarek Heiba. The researcher will bear ultimate responsibility for all activities associated with the conduct of a research project including recruitment of patients, explaining and performing the procedures to them,A total of 40 volunteer patients with at least 2 non-cavitated molar teeth will be assigned in this study. Patients will be randomly divided into two groups according to type of sealant (S) where in group S1, pits and fissures will be sealed with bioactive pits-and-fissure sealant; while group S2, pits and fissures will be sealed with fluoride releasing resin based pits and fissures sealant. Each restoration will be assessed after three, six months,The tooth will be illuminated with a violet light approximately 405 nm thus stimulating both prophyrins to emit red light that contains less energy. the denser the bacteria colonization on tooth's surface, the more intense the red fluorescent signal; in contrast sound enamel sent out a green fluorescent signal. These light signals are recorded by the highly developed optics and analyzed by the device's software. The software filters and quantifies the fluorescence emitted by the dental tissue and converts the relationship between green and red.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be 16-25 Years old
* Patient should have good oral hygiene and general health with at least 2 •sound intact occlusal surfaces of first and/or second molar teeth in each quadrant of maxilla or mandible.

Exclusion Criteria:

* Known allergy to any of the resins used
* Clinically detectable caries
* Previously placed sealants or restorations
* Bruxism or malocclusion

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
caries incidence | six months
  development of pit and fissure caries

IPD SHARING:
Plan to Share IPD: Undecided